CLINICAL TRIAL: NCT00324740
Title: A Phase I/II Study of Vorinostat (Suberoylanilide Hydroxamic Acid, SAHA) in Combination With Isotretinoin (13-cis Retinoic Acid, 13-CRA) in the Treatment of Patients With Advanced Renal Cell Carcinoma
Brief Title: Vorinostat and Isotretinoin in Treating Patients With Advanced Kidney Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00095; NCI-2009-00095 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-6896 (Other: NCI/CTEP); N01CM62204 (NIH); P30CA013330 (NIH)
Record Dates: First submitted 2006-05-10; First posted 2006-05-11 (Estimated); Results first posted 2015-11-24 (Estimated); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Recurrent Renal Cell Cancer; Stage III Renal Cell Cancer; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Vorinostat; Isotretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (vorinostat and isotretinoin) (Experimental): Patients receive oral vorinostat (SAHA) twice daily and oral isotretinoin twice daily on days 3-5, 10-12, 17-19, and 24-26. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: vorinostat; Drug: isotretinoin

INTERVENTIONS:
Drug: vorinostat — Given orally
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Drug: isotretinoin — Given orally
  Other Names: 13-CRA; Amnesteem; Cistane; Claravis; Sotret

SUMMARY:
This phase I/II trial is studying the side effects and best dose of isotretinoin when given together with vorinostat and to see how well they work in treating patients with advanced kidney cancer. Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Isotretinoin may cause kidney cancer cells to look more like normal cells, and to grow and spread more slowly. Giving vorinostat together with isotretinoin may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose and phase II dose of isotretinoin when given in combination with vorinostat (SAHA) in patients with advanced renal cell carcinoma. (Phase I) II. Define dose-limiting and other toxicities in patients treated with this regimen. (Phase I) III. Determine the objective response rate of patients treated with this regimen. (Phase II)

SECONDARY OBJECTIVES:

I. Conduct a pharmacokinetic analysis of this regimen in these patients. (Phase I) II. Conduct gene profiling analysis of pre-study, paraffin-embedded tissues from patients treated with this regimen. (Phase I) III. Conduct correlative studies to identify the effect of SAHA and isotretinoin on RAR-B, LRAT, and STAT1-3 expression. (Phase I)

OUTLINE: This is a multicenter, phase I, dose-escalation study of isotretinoin, followed by a multicenter, phase II, prospective, non-randomized study.

Phase I: Patients receive oral vorinostat (SAHA) twice daily and oral isotretinoin twice daily on days 3-5, 10-12, 17-19, and 24-26. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of isotretinoin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

Phase II: Patients receive SAHA as in phase I and isotretinoin as in phase I at the MTD determined in phase I. Tissue and blood samples are obtained for biomarker/laboratory studies in weeks 1 and 4.

Gene profile analysis is conducted on tumor tissue. After completion of study treatment, patients are followed for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed renal cell carcinoma

  * Advanced or metastatic disease
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion > 20 mm by conventional techniques or > 10 mm by spiral CT scan (phase II only)
* Failed ≥ 2 prior treatment regimens, including chemotherapy, immunotherapy (i.e., interleukin or interferon), biological agents (i.e., kinase inhibitors), or combinations thereof

  * An overlap between classes of therapies given concurrently will be counted as 2 prior treatment regimens
* No known brain metastases
* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Life expectancy > 3 months
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.5 mg/dL
* AST and ALT < 2.5 times upper limit of normal
* Creatinine ≤ 2 mg/dL OR creatinine clearance > 50 mL/min
* Negative pregnancy test

Exclusion criteria:

* Not pregnant or nursing
* No history of allergic reactions or hypersensitivity attributed to compounds of similar chemical or biologic composition to vorinostat (SAHA), isotretinoin, or other agents or components (e.g., parabens) used in this study
* No uncontrolled intercurrent illness, including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situation that would preclude study compliance
* No concurrent antiretroviral therapy for HIV-positive patients
* No other concurrent anticancer therapy, including radiation, biologic, or chemotherapeutic agents, for renal cell carcinoma or other tumors
* No other concurrent investigational agents, valproic acid, or other retinoid

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-03; Primary Completion 2011-02 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Nanus, Principal Investigator — Montefiore Medical Center - Moses Campus
Locations (2):
- United States (2):
  - Weill Medical College of Cornell University, New York, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 14 patients were enrolled between June 2006 and September 2010
Groups:
- Dose Level 1: Vorinostat (300mg) and Isotretinoin (0.25 mg/kg): Patients receive oral vorinostat (SAHA-300 mg) twice daily and oral isotretinoin (0.25 mg/kg) twice daily for 3 consecutive days per week (Tues/Wed/Thurs). Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  vorinostat: Given orally
  isotretinoin: Given orally
- Dose Level 2 Vorinostat (300mg) and Isotretinoin (0.375 mg/kg): Patients receive oral vorinostat (SAHA-300 mg) twice daily and oral isotretinoin (0.375 mg/kg) twice daily for 3 consecutive days per week (Tues/Wed/Thurs). Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  vorinostat: Given orally
  isotretinoin: Given orally
- Dose Level 3: Vorinostat (300mg) and Isotretinoin (0.5 mg/kg): Patients receive oral vorinostat (SAHA-300 mg) twice daily and oral isotretinoin (0.5 mg/kg) twice daily for 3 consecutive days per week (Tues/Wed/Thurs). Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  vorinostat: Given orally
  isotretinoin: Given orally
Period: Overall Study
Arm/Group | Dose Level 1: Vorinostat (300mg) and Isotretinoin (0.25 mg/kg) | Dose Level 2 Vorinostat (300mg) and Isotretinoin (0.375 mg/kg) | Dose Level 3: Vorinostat (300mg) and Isotretinoin (0.5 mg/kg)
Started | 7 | 3 | 4
Completed | 6 | 3 | 3
Not Completed | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Vorinostat and Isotretinoin)
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 55 [33 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 3
Race/Ethnicity, Customized [Number; unit: participants]
  White | 6
  Asian | 1
  Black | 1
  Native Hawaiin or other Pacific Islander | 1
  Unknown | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Dose Limiting Toxicity Associated With Vorinostat Concurrently Administered With Isotretinoin
Description: Defined as the occurrence of one or more of the following toxicities as graded by the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0
Time Frame: Course 1, up to 28 days
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 1: Vorinostat (300mg) and Isotretinoin (0.25 mg/kg); Dose Level 2 Vorinostat (300mg)and Isotretinoin (0.375 mg/kg); Dose Level 2 Vorinostat (300mg)and Isotretinoin (0.5 mg/kg): Patients receive oral vorinostat (SAHA) and oral isotretinoin twice daily for 3 consecutive days per week (Tues/Wed/Thurs). Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  vorinostat: Given orally
  isotretinoin: Given orally
Arm/Group | Dose Level 1: Vorinostat (300mg) and Isotretinoin (0.25 mg/kg) | Dose Level 2 Vorinostat (300mg)and Isotretinoin (0.375 mg/kg) | Dose Level 2 Vorinostat (300mg)and Isotretinoin (0.5 mg/kg)
Number analyzed (Participants) | 6 | 3 | 3
Participants | 1 | 0 | 0

2. Primary Outcome: Maximum Tolerated Dose of Vorinostat in Combination With Isotretinoin
Description: Hematologic: Any Grade 3/4 Thrombocytopenia and/or Grade 3/4 Neutropenia Non-Hematologic: Any >/= Grade3 non-hematologic toxicity considered by the investigator to be possibly related to study drug and/or any non-hematologic toxicity that results in a dose-delay of more than three weeks.
Time Frame: Once 2 DLT events occur in patients, the preceding dose will be designated the maximum tolerated dose (MTD).
Population: The recommended phase II dose is vorinostat (300 mg bid) + Isotretinoin (0.5 mg/kg PO bid) three days per week
Measure: Number; unit: mg/kg BID
Arm/Group | Treatment (Vorinostat and Isotretinoin)
Number analyzed (Participants) | 12
mg/kg BID | 0.5

3. Primary Outcome: Objective Response Rate
Description: The Response Evaluation Criteria in Solid Tumors (RECIST 1.0) was used and tumor responses were defined as complete response (CR), partial response (PR), stable disease (SD) or Progression
Time Frame: Tumor measurements every 8 weeks until disease progression
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: Vorinostat (300mg) and Isotretinoin (0.25 mg/kg) | Dose Level 2 Vorinostat (300mg)and Isotretinoin (0.375 mg/kg) | Dose Level 2 Vorinostat (300mg)and Isotretinoin (0.5 mg/kg)
Number analyzed (Participants) | 5 | 3 | 3
Participants
  Partial Response | 0 | 1 | 0
  Stable Disease | 4 | 2 | 3
  Progression | 1 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Treatment (Vorinostat and Isotretinoin)
Serious Adverse Events (participants affected / at risk) | 11/12
Other Adverse Events (participants affected / at risk) | 4/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Vorinostat and Isotretinoin) (N=12)
Fatigue (General disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
Anxiety (Nervous system disorders) | 1 (1)
Depression (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Vorinostat and Isotretinoin) (N=12)
Weight Loss (General disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less